CLINICAL TRIAL: NCT06906653
Title: Population Health Management for Kaiser Permanente Northern California (KPNC) Members With Newly Diagnosed Diabetes: A Randomized Trial of a Proactive and Augmented Initial Care Strategy
Brief Title: Population Health Management for KPNC Members With Newly Diagnosed Diabetes: A Randomized Trial of a Proactive and Augmented Initial Care Strategy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: The Permanente Medical Group (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2220224
Record Dates: First submitted 2025-03-24; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes; Type 2 Diabetes Mellitus (T2DM); Type 2 Diabetes (T2D)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Initial Type 2 Diabetes (T2D) Care (No Intervention): Patients in the usual care arm will receive the standard T2D care provided to Kaiser Permanente Northern California members with recently diagnosed T2D. This care includes any counseling or treatment recommendations made by the primary care provider and the assigned care manager.
- Augmented Initial Type 2 Diabetes (T2D) Care (Experimental): The intervention - Augmented Initial T2D Care - comprises the elements of usual care augmented by more proactive and intensive outreach from the diabetes care team and self-management support by care managers, health educators, and dieticians.
  Interventions: Behavioral: Augmented Initial Type 2 Diabetes Care

INTERVENTIONS:
Behavioral: Augmented Initial Type 2 Diabetes Care — The intervention will include 4 components: 1) Making primary care providers (PCPs) aware that the patient has been selected to receive "Augmented Initial Type 2 Diabetes (T2D) Care", 2) encouraging early care manager outreach to establish care, ensure prescribing of appropriate medications, and support medication adherence, 3) a one-on-one virtual health educator visit to reinforce self-management education and ensure set-up of remote glucose monitoring or continuous glucose monitoring (if eligible), and 4) a one-on-one virtual nutrition visit to provide individualized counseling.
  Arms: Augmented Initial Type 2 Diabetes (T2D) Care

SUMMARY:
This study is a 2-arm randomized trial of Augmented Initial Type 2 Diabetes (T2D) Care vs. Usual Initial T2D Care among adults (18-74 years) with newly diagnosed T2D who have risk factors (defined by age and diagnosis HbA1c value) for suboptimal early glycemic control. Augmented Initial T2D Care comprises the elements of usual care augmented by more proactive and intensive outreach from the diabetes care team. The study team will use electronic health record (EHR) data to assess between-arm differences in diabetes-related outcomes at 6- and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-74 years
* Newly diagnosed with type 2 diabetes
* Kaiser Permanente Northern California member receiving care in a participating service area
* If age ≤45 years, then HbA1c>8%
* If age<45 years, then HbA1c>10%

Exclusion Criteria:

* Individuals who are pregnant
* Individuals with likely type 1 diabetes (T1D)

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Average hemoglobin A1c (HbA1c) | 6-months
  Between-arm differences in HbA1c
Average hemoglobin A1c (HbA1c) | 12-months
  Between-arm differences in HbA1c

SECONDARY OUTCOMES:
Time to achievement of glycemic targets | 6-months
Time to achievement of glycemic targets | 12-months
Adherence to HbA1c monitoring | 6-months
  Number of participants with a new HbA1c laboratory value
Adherence to HbA1c monitoring | 12-months
  Number of participants with a new HbA1c laboratory value
Type 2 diabetes medication and statin initiation | 6-months
  Number of participants who are prescribed a type 2 diabetes medication and/or statin
Type 2 diabetes medication and statin initiation | 12-months
  Number of participants who are prescribed a type 2 diabetes medication and/or statin
Type 2 diabetes medication adherence | 6-months
  Proportion of days covered since initiation
Type 2 diabetes medication adherence | 12-months
  Proportion of days covered since initiation
Completion of preventative screening | 6-months
  Number of participants who complete retinal and microalbuminuria screening
Completion of preventative screening | 12-months
  Number of participants who complete retinal and microalbuminuria screening

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente Division of Research, Pleasanton, California, United States

IPD SHARING:
Plan to Share IPD: No